CLINICAL TRIAL: NCT05220865
Title: Hall Technique or Modified Hall Technique of Deep Carious Lesions in Primary Molars: A Randomized Clinical Trial
Brief Title: Hall Technique or Modified Hall Technique of Deep Carious Lesions in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, AYŞE IŞIL CİHAN, Professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2-21-956
Record Dates: First submitted 2022-01-22; First posted 2022-02-02 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Dental Caries in Children; Tooth Diseases; Tooth Demineralization; Stomatognathic Diseases
Keywords: Hall Technique; Deep dentine caries; Carious primary molars
MeSH Terms: conditions — Tooth Diseases; Tooth Demineralization; Stomatognathic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, investigator evaluating treatment success at follow-up appointments and biostatistician will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hall Technique (Active Comparator): A preformed metal crown will be cemented on the carious primary molar tooth without any tooth preparation and local anesthesia.
  Interventions: Procedure: Hall Technique
- Modified Hall Technique (Experimental): In the Modified Hall technique only infected soft dentin tissue will be removed with hand instruments and a preformed metal crown will be placed with Hall technique.
  Interventions: Procedure: Modified Hall Technique

INTERVENTIONS:
Procedure: Hall Technique — * Only food scraps or debris will be removed from the caries cavity.
  * The smallest crown size will be selected that covers all cusps and approaches the contact points with a slight "springback" feel.
  * If the contact points are tight, orthodontic elastic separators will be placed through the contacts and the SSC will be placed at the second appointment 3-5 days later.
  * The SSC will be loaded with glass ionomer luting cement and placed evenly on the tooth.
  * The child will be asked to bite firmly until the crown is pushed down over the tooth.
  * If the child is unable or unwilling to bite down on the SSC, finger pressure will be used to seat the crown
  * The child will continue to bite on a cotton roll until the cement hardens
  * Excess glass ionomer cement will be removed from the crown margins with hand instruments and dental floss.
  Arms: Hall Technique
Procedure: Modified Hall Technique — * Food scraps or debris will be cleaned from the caries cavity and infected soft carious dentin tissue will be excavated with hand instruments.
  * The smallest crown size will be selected that covers all cusps and approaches the contact points with a slight "springback" feel.
  * If the contact points are tight, orthodontic elastic separators will be placed through the contacts and the SSC will be placed at the second appointment 3-5 days later.
  * The SSC will be loaded with glass ionomer luting cement and placed evenly on the tooth.
  * The child will be asked to bite firmly until the crown is pushed down over the tooth.
  * If the child is unable or unwilling to bite down on the SSC, finger pressure will be used to seat the crown
  * The child will continue to bite on a cotton roll until the cement hardens
  * Excess glass ionomer cement will be removed from the crown margins with hand instruments and dental floss.
  Arms: Modified Hall Technique

SUMMARY:
The purpose of this randomized clinical trial is to compare the clinical/radiographic success of Hall technique and modified Hall technique in the treatment of primary molars with deep dentine carious lesions in children (3-12-year-old). The secondary aim is to examine the effect of marginal ridge breakdown level on treatment success.

DETAILED DESCRIPTION:
Untreated caries in deciduous teeth affect 532 million children worldwide. According to the Turkey Oral and Dental Health Profile study conducted in 2018, the prevalence of untreated caries in 5-year-old children is 64.4%. The traditional treatment of dentine caries is to restore the teeth after removal of the carious tissue. There is increasing evidence for minimally invasive interventions as an alternative to this traditional operative/restorative treatment.

One of the minimally invasive treatment approaches applied in children is the Hall Technique. Local anesthesia and tooth preparation are not required in this technique, and decayed primary molars are covered with stainless steel crowns without removing any carious tissue. The Hall technique has advantages such as preventing aerosol formation, shortening the treatment time, increasing patient cooperation, and reducing the need for general anesthesia and sedation in noncompliant patients. Its popularity has also increased during the Covid-19 process.

The success of the Hall technique in primary teeth with deep caries has been investigated in a limited number of clinical studies, and it has been observed that the technique has lower success rates in teeth with deep caries than in teeth with shallow/medium depth caries. To answer the question of whether modifying the Hall technique (removing the necrotic carious dentin layer manually with excavators before placing a stainless-steel crown) in deeply carious primary molars will increase the success of the original Hall technique (placing stainless steel crown without any intervention to the carious lesion), a randomized study was designed.

268 healthy children between the ages of 3-12 will be recruited from Ankara Yıldırım Beyazıt University Faculty of Dentistry, Department of Pediatric Dentistry outpatient clinic. Participants who met the inclusion criteria and agreed to participate will be randomly allocated to Group 1 (Modified Hall Technique) or Group 2 (Hall Technique).

The allocation of patients in each group will be carried out by a random list. The sequence will be generated by a computerized random number generator. Enclosed assignments in sequentially numbered, opaque, sealed envelopes will be used as allocation concealment mechanism. Group allocation will be performed by an independent researcher, not involved in the study.

Clinical and radiographic success of treatments will be determined at follow-up appointments at 3rd, 6th and 12th months by one blinded examiner. In follow-up appointments; treatments will be recorded as "successful" (restoration appears satisfactory, no intervention required/ no clinical signs or symptoms of pulpal pathology/ no pathology visible on radiographs/ tooth exfoliated), "minor failure" (crown perforation/ new caries (around margins)/ restoration loss; tooth restorable/ reversible pulpitis treated without requiring pulpotomy or extraction) or "major failure" (irreversible pulpitis or dental abscess requiring pulpotomy or extraction/ inter-radicular radiolucency/ restoration loss; tooth unrestorable/ internal root resorption).

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy children
* Participants attending follow-up appointments
* Children having at least one primary molar tooth with deep dentin caries involving occluso proximal surfaces.

Tooth inclusion criteria:

* Vital pulp with symptom-free or reversible pulpitis
* Presence of marginal ridge breakdown and accessible cavity with hand instruments,
* Presence of active cavitated carious lesion (Code 3 with Nyvad criteria for caries lesion activity and severity assessment- Nyvad et al., 1999)
* Absence of spontaneous or prolonged pain related with irreversible pulpitis
* Absence of fistula or abscess near the tooth
* Absence of pathological mobility
* Absence of pain on percussion
* Absence of pulp exposure
* Caries lesion located in ½ inner part of dentin radiographically
* Presence of sound dentin layer between the deepest part of the carious lesion and the pulp radiographically
* Absence of periapical or furcation pathologies on radiographs
* Absence of internal and external root resorption on radiographs
* More than ½ of root remaining

Exclusion Criteria:

* Any systemic disease, physical or mental disorder
* Children or parents who doesn't accept to participate and sign the informed consent
* Clinical or radiographic signs of pulpal or peri-radicular pathology
* Caries cavity which cannot be accessible to hand instruments
* Physiological root resorption more than 1/2 of the root in primary molars

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 268 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical and radiographic success of the treatments | Change from baseline up to 3, 6 and 12 months
  The clinical evaluation will be performed by one blinded examiner with the criteria as proposed by Innes et al. (2007).
  Outcome criteria for the clinical and radiographic assessment of restorations and teeth will be as follows:
  Treatments will be considered as "successful" if the restoration appears satisfactory (no intervention required), no clinical signs or symptoms of pulpal pathology, no pathology visible on radiographs or tooth exfoliated
  The treatments will be classified as "minor failure" if there is a crown perforation, new caries around margins, restoration loss (tooth restorable) and/or reversible pulpitis treated without requiring pulpotomy or extraction.
  The treatments will be classified as "major failure" if there is irreversible pulpitis or dental abscess requiring pulpotomy or extraction, inter-radicular radiolucency, restoration loss (tooth unrestorable) and/or internal root resorption (Innes et al., 2007).

SECONDARY OUTCOMES:
The effect of the amount of marginal ridge fracture on treatment success | Change from baseline up to 3, 6 and 12 months
  The extent of marginal ridge breakdown will be determined by the ratio of the amount of fractured marginal ridge to the total marginal ridge of the tooth and will be scored in 4 groups (<25%, 25-50%, 50-75%, >75%) (Cho et al.,2018).

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe I. Orhan, Assoc. Prof., Study Chair — Ankara Yıldırım Beyazit University Faculty of Dentistry
Locations (1):
- Ankara Yıldırım Beyazıt University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boyd DH, Thomson WM, Leon de la Barra S, Fuge KN, van den Heever R, Butler BM, Leov F, Foster Page LA. A Primary Care Randomized Controlled Trial of Hall and Conventional Restorative Techniques. JDR Clin Trans Res. 2021 Apr;6(2):205-212. doi: 10.1177/2380084420933154. Epub 2020 Jun 19. PMID 32559403
- [Background] Boyd DH, Page LF, Thomson WM. The Hall Technique and conventional restorative treatment in New Zealand children's primary oral health care - clinical outcomes at two years. Int J Paediatr Dent. 2018 Mar;28(2):180-188. doi: 10.1111/ipd.12324. Epub 2017 Aug 8. PMID 28787534
- [Background] Eden E, Frencken J, Gao S, Horst JA, Innes N. Managing dental caries against the backdrop of COVID-19: approaches to reduce aerosol generation. Br Dent J. 2020 Oct;229(7):411-416. doi: 10.1038/s41415-020-2153-y. Epub 2020 Oct 9. PMID 33037360
- [Background] GBD 2017 Oral Disorders Collaborators; Bernabe E, Marcenes W, Hernandez CR, Bailey J, Abreu LG, Alipour V, Amini S, Arabloo J, Arefi Z, Arora A, Ayanore MA, Barnighausen TW, Bijani A, Cho DY, Chu DT, Crowe CS, Demoz GT, Demsie DG, Dibaji Forooshani ZS, Du M, El Tantawi M, Fischer F, Folayan MO, Futran ND, Geramo YCD, Haj-Mirzaian A, Hariyani N, Hasanzadeh A, Hassanipour S, Hay SI, Hole MK, Hostiuc S, Ilic MD, James SL, Kalhor R, Kemmer L, Keramati M, Khader YS, Kisa S, Kisa A, Koyanagi A, Lalloo R, Le Nguyen Q, London SD, Manohar ND, Massenburg BB, Mathur MR, Meles HG, Mestrovic T, Mohammadian-Hafshejani A, Mohammadpourhodki R, Mokdad AH, Morrison SD, Nazari J, Nguyen TH, Nguyen CT, Nixon MR, Olagunju TO, Pakshir K, Pathak M, Rabiee N, Rafiei A, Ramezanzadeh K, Rios-Blancas MJ, Roro EM, Sabour S, Samy AM, Sawhney M, Schwendicke F, Shaahmadi F, Shaikh MA, Stein C, Tovani-Palone MR, Tran BX, Unnikrishnan B, Vu GT, Vukovic A, Warouw TSS, Zaidi Z, Zhang ZJ, Kassebaum NJ. Global, Regional, and National Levels and Trends in Burden of Oral Conditions from 1990 to 2017: A Systematic Analysis for the Global Burden of Disease 2017 Study. J Dent Res. 2020 Apr;99(4):362-373. doi: 10.1177/0022034520908533. Epub 2020 Mar 2. PMID 32122215
- [Background] Innes NP, Stirrups DR, Evans DJ, Hall N, Leggate M. A novel technique using preformed metal crowns for managing carious primary molars in general practice - a retrospective analysis. Br Dent J. 2006 Apr 22;200(8):451-4; discussion 444. doi: 10.1038/sj.bdj.4813466. PMID 16703041
- [Background] Innes NP, Evans DJ, Stirrups DR. The Hall Technique; a randomized controlled clinical trial of a novel method of managing carious primary molars in general dental practice: acceptability of the technique and outcomes at 23 months. BMC Oral Health. 2007 Dec 20;7:18. doi: 10.1186/1472-6831-7-18. PMID 18096042
- [Background] Nyvad B, Baelum V. Nyvad Criteria for Caries Lesion Activity and Severity Assessment: A Validated Approach for Clinical Management and Research. Caries Res. 2018;52(5):397-405. doi: 10.1159/000480522. Epub 2018 Mar 5. PMID 29506010
- [Derived] Konukman Turker S, Cihan AI. Two-year outcomes of hall technique and modified hall technique in deep carious lesions of primary molars: a randomized clinical trial. BMC Oral Health. 2026 Jan 12. doi: 10.1186/s12903-026-07667-2. Online ahead of print. PMID 41526924
- See also: Cho V, Anthonappa R, King N." Marginal Ridge Breakdown as a Predictor for Pulpal Involvement in Primary Molar". The International Association of Pediatric Dentistry. Global Summit on Early Childhood Caries. — https://program.eventact.com/viewabstract?Abst=182712&Code=3855981